CLINICAL TRIAL: NCT00258570
Title: Genetic Polymorphisms in Idiopathic Pulmonary Fibrosis
Brief Title: Genetic Polymorphisms in Idiopathic Pulmonary Fibrosis (IPF)
Acronym: GP
Status: Recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Kevin F. Gibson, Professor of Medicine, University of Pittsburgh
Other Study IDs: STUDY20030223
Record Dates: First submitted 2005-11-23; First posted 2005-11-24 (Estimated); Last update posted 2025-11-12 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Fibrosis
Keywords: "Lung[A04.400]"
MeSH Terms: conditions — Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood samples retained for multitude of testing. Consent allows for unrestricted use of samples.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purposes of this study are:

* to determine if there are specific genetic traits that might explain why patients have developed pulmonary fibrosis;
* to determine if specific genetic traits account for differing patterns of inflammation and scar tissue that has formed in the patient's lungs.

DETAILED DESCRIPTION:
Idiopathic pulmonary fibrosis (IPF) is a disease of unknown etiology that is characterized by the insidious development of lung fibrosis ultimately leading to distortion of the lung architecture, respiratory failure, and death. IPF is one of several entities associated with pulmonary fibrosis called the idiopathic interstitial pneumonias (IIP). Based on the histopathologic features of the fibrotic process, it is possible to identify four distinct entities: usual interstitial pneumonia (UIP) (synonymous with IPF), nonspecific interstitial pneumonia (NSIP), desquamative interstitial pneumonia DIP), and acute interstitial pneumonia (AIP) (Hamman-Rich lung). Each type appears to have different clinical progression and a different response to anti-inflammatory therapy. Our overall objective is to elucidate the molecular pathogenesis of IPF (UIP) by identifying factors that determine host susceptibility to this disease. We hypothesize that patients who develop pulmonary fibrosis, have a genetic propensity to abnormal lung repair that leads to fibrosis after acute lung injury. We further hypothesize that these genetic susceptibilities may determine if the pathologic process in the lung after an insult becomes UIP, AIP, NSIP, or DIP. To explore these hypotheses we propose to characterize the genetic polymorphisms in candidate genes involved in inflammation, matrix turnover, fibroblast proliferation and differentiation, and epithelial cell proliferation; and to correlate this with indices of disease progression.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Diagnosis of pulmonary fibrosis confirmed by physical examination, pulmonary function testing, chest X-ray, and computed tomography (CT) scans.
* Adult patients who are seeking treatment at the Dorothy P. and Richard P. Simmons Center for Interstitial Lung Disease.

Exclusion Criteria:

* Under 18 years of age
* Non-fibrotic ILD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient population includes patients who have been diagnosed with a fibrotic interstitial lung disease who have been seen by a Simmons Center Physician.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2003-01; Primary Completion 2035-07 (Estimated); Study Completion 2035-07 (Estimated)

PRIMARY OUTCOMES:
Genetic Polymorphisms in Idiopathic Pulmonary Fibrosis (IPF) | Sample collection will occur up to 5 years based on the current rate of sample collection.
  Blood samples will be collected to validate in a large cohort the per- allele associations of prespecified SNPs with IPF case status adjusted for age , sex. smoking, and principal components of ancestry.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin F Gibson, MD, Principal Investigator — University of Pittsburgh, Simmons Center for ILD
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- See also: The Dorothy P. and Richard P. Simmons Center for Interstitial Lung Disease is designed to provide patient-friendly advice and support for people with idiopathic pulmonary fibrosis. — http://www.upmc.com/services/pulmonology/interstitial-lung-disease/